CLINICAL TRIAL: NCT04993599
Title: Evaluation of Social Robot Usability for Pediatric Patients and Carers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-05-085-006
Record Dates: First submitted 2021-07-16; First posted 2021-08-06 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-07

CONDITIONS: Pediatrics
Keywords: Pediatrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric patients (Experimental): <Intervention> The participants(Pediatric patients) mainly interact with the social robot which is controlled by the researcher behind the scene
  Interventions: Device: Social robot interaction
- Carers (Experimental): <Intervention> The participants(Carers) interact with the social robot and watch how their child interact with the robot which is controlled by the researcher behind the scene
  Interventions: Device: Social robot interaction

INTERVENTIONS:
Device: Social robot interaction — The participants interact with the social robot which is controlled by the researcher behind the scene (wizard of oz. method).

SUMMARY:
This study is conducted for a mixed methods study. Subjects are 20 child patients and 20 their carers. First, Participants use and interact with a social robot. The robot is controlled by researcher with the wizard of oz. method. The interaction is video-recorded for the later analysis of the child's engagement through amount of his vocalization and sentences. After using social robot, a survey and an in-depth interview will be done.

This study investigates the usability, satisfaction, emotion, and other dimensions of social robots of pediatric patients and carers and evaluate the degree of interaction with them with the recording data, survey and in-depth interview. This study is a basis for using social robots to pediatric patients in the hospital environments.

DETAILED DESCRIPTION:
This study is conducted for a mixed methods study. Subjects are 20 child patients and 20 their carers. First, Participants use and interact with a social robot. The robot is controlled by researcher with the wizard of oz. method. And another researcher observes the participants-robot interaction. The interaction is video-recorded for the later analysis of the child's engagement through amount of his vocalization and sentences. After using social robot, a survey and an in-depth interview will be done.

This study investigates the usability, satisfaction, emotion, and other dimensions of social robots of pediatric patients and carers and evaluate the degree of interaction with them with the recording data, survey and in-depth interview. This study is a basis for using social robots to pediatric patients in the hospital environments.

ELIGIBILITY:
<Pediatric patients>

Inclusion Criteria:

* Patients visiting Samsung Medical Center (Age 5~12)
* A person who voluntarily agrees to participate in the study
* Patients who are able to agree with a consent

Exclusion Criteria:

* Those who disagree with the study
* Patients and carers who find it difficult to interact with the robot

<Carers>

Inclusion Criteria:

* Caregivers of the patient participant
* Adults over 19 years of age
* A person who voluntarily agrees to participate in the study

Exclusion Criteria:

* Those who disagree with the study
* Patients and carers who find it difficult to interact with the robot

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Duration and time of robot communication with the participants | Through study completion, an average of 1 year
  Assessment of how long the duration and time of the communication between the participants ans robot is.
Number of conversations exchanged between the participant and the robot | Through study completion, an average of 1 year
  Assessment of the number of conversations exchanged between the participant and the robot
The amount of the incidence of participants' vocalization when interacting with the robot | Through study completion, an average of 1 year
  Assessment of the incidence of participants' vocalization when interacting with the robot.

SECONDARY OUTCOMES:
A qualitative study on user experience | Through study completion, an average of 1 year
  A qualitative study on user experience using a in-depth interview
A quantitative study on the user experience | Through study completion, an average of 1 year
  A quantitative study on the user experience using User Experience Questionnaire. The items have the form of a semantic differential, i.e. each item is represented by two terms with opposite meanings. The items are scaled from -3 to +3. Thus, -3 represents the most negative answer, 0 a neutral answer, and +3 the most positive answer.

CONTACTS AND LOCATIONS:
Overall Officials: Meong Hi Son, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Centre, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided